CLINICAL TRIAL: NCT00590837
Title: Randomized Prospective Study of Adding Lomustine to Idarubicin and Cytarabine for Induction and Post-remission Chemotherapy in Older Patients With Acute Myeloid Leukaemia, and Feasibility of Allogeneic Transplantation for Patients From 60 to 65 Years Old
Brief Title: Adding Lomustine to Chemotherapy in Older Patients With Acute Myelogenous Leukemia (AML), and Allogeneic Transplantation for Patients From 60 to 65 Years Old
Acronym: LAM-SA 2007
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2007/13
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Chemotherapy; older; De novo AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients will be treated by adding lomustine to chemotherapy
  Interventions: Drug: Lomustine
- 2 (No Intervention): Patients will be treated without adding lomustine to chemotherapy

INTERVENTIONS:
Drug: Lomustine — Induction: chemotherapy + lomustine (CCNU), 200 mg/m2 orally at day 1.
  Consolidation: chemotherapy + lomustine (CCNU), 80 mg orally at day 1.
  Reinductions: chemotherapy + lomustine (CCNU), 40 mg orally at day 1.
  Arms: 1

SUMMARY:
A multicenter randomized trial comparing induction therapy (IC: Idarubicin and Cytarabine, 5 + 7) to ICL (the same drugs plus lomustine (CCNU), 200 mg/m2 orally at day 1). Patients in complete remission (CR) will then receive a post-remission schedule with or without lomustine according to randomization. Patients from 60 to 65 years old will be proposed to reduced conditioning allogeneic transplantation after first consolidation.

DETAILED DESCRIPTION:
* Principal Objective: The primary objective of this study is to assess the ability of lomustine to increase the overall survival by adding lomustine to induction and post-remission chemotherapy.
* Secondary Objectives:

  * To assess the ability of lomustine to increase the CR rate.
  * To assess the ability of lomustine to increase the event-free survival.
  * To evaluate the toxicity and side-effects of lomustine.
  * To evaluate the feasibility of reduced conditioning allogeneic transplantation *between 60 and 65 years old.
  * To evaluate prognostic factors.
  * To evaluate QOL in elderly.
* Study design: Parallel
* Study plan:

  * Induction therapy: Patients will be randomized to receive idarubicin (5d) plus cytarabine or the same drugs plus lomustine, the latter given at the dose of 200 mg/m2 orally at day 1.
  * Consolidation therapy: After completing induction treatment, patients who are in complete remission will receive a course of consolidation therapy with idarubicin (3d) and subcutaneous cytarabine.
  * Maintenance therapy: In all patients with persisting CR one month after completing consolidation: six courses of monthly combination chemotherapy (idarubicin (1d) and subcutaneous cytarabine) and then a continuous regimen of methotrexate and 6-mercaptopurine, for 6 months.
  * Allogeneic transplantation: Patients between 60 and 65 years old with a full matched donor will receive after consolidation (if still in CR) an alloBMT with a reduced conditioning regimen of Fludarabine (3d) and TBI (2Gy).
* Number of subjects: 460

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years and older with de novo AML and non-poor cytogenetic features.
* Patients with no unfavourable cytogenetic (based on GOELAMS-BGMT criteria)
* Performance status and Sorror score < 3 .
* Signed and dated informed consent.

Exclusion Criteria:

* Acute promyelocytic leukemia.
* Patients with myeloproliferative syndromes prior to diagnosis of AML.
* Patients who previously had myelodysplastic syndrome.
* Positive serology for HIV.
* Patients with unfavourable cytogenetic
* Patients with an isolated medullary extra localization of their disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 year

SECONDARY OUTCOMES:
Complete remission | 1 year
Event-free survival | 1 year
Prognostic factors | 1 year
Quality of Life (QOL) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Pigneux, MD, PhD, Principal Investigator — University Hospital Bordeaux, France
Locations (32):
- France (32):
  - Services maladies du sang, cancérologie, Hôpital Sud, CHU Amiens, Amiens
  - Service des maladies du sang, Centre Hospitalier Universitaire d'Angers, Angers
  - Service Hématologie, Centre Hospitalier Annecy, Annecy
  - C.H Victor Dupouy, Argenteuil
  - Service Médecine Interne, Onco-Hématologie, Maladies Infectieuses, Hôpital Henri Duffaut, Centre Hospitalier Avignon, Avignon
  - Service Hématologie, Centre Hospitalier de la Côte Basque, Bayonne
  - Service Hématologie, Hôpital Minjoz, Besançon
  - Unité Hématologie, Centre Hospitalier Blois, Blois
  - Service des maladies du sang - Hôpital Haut-Lévêque, Bordeaux - Pessac
  - Service Hématologie, Hôpital Dr Duchenne, Boulogne-sur-Mer
  - Service Hématologie, Hôpital Augustin Morvan, Brest
  - Service Hématologie et Thérapie cellulaire, Pavillon Villemin Pasteur, CHU Clermont-Ferrand, Clermont-Ferrand
  - Service Oncologie - Hématologie, Hôpital Pasteur, Centre Hospitalier Colmar, Colmar
  - Service Hématologie Clinique, CHU Dijon Hôpital des enfants, Dijon
  - Service Hématologie Clinique, Hôpital Michallon, CHU de Grenoble, Grenoble
  - Service Onco-Hématologie 3, Institut Paoli Calmettes, Marseille
  - Service Hématologie Oncologie, CHR Metz-Thionville, Metz
  - Service Hématologie Oncologie, Hôpital Lapeyronie, CHU de Montpellier, Montpellier
  - Département d'hématologie, Hôpital E.Muller, Centre Hospitalier de Mulhouse, Mulhouse
  - Service Hématologie Clinique, CHU -Hôtel Dieu, Nantes
  - Service Hématologie Clinique, Hôpital Archet 1, Nice
  - Service Médecine B - Unité Onco-hématologique, CHU Caremeau, Nîmes
  - Service Oncologie Médicale, Hôpital de la Source, Orléans
  - Unité d'Hématologie, Hôpital Cochin, Paris
  - Service Hématologie, CHG Saint Jean, Perpignan
  - Service Hématologie Clinique, Hôpital Robert Debre, Reims
  - Service Hématologie Clinique, Hôpital Pontchaillou, Rennes
  - Service d'Hématologie, Institut de Cancérologhie de la Loire, Saint Priez En Jarez
  - Département d'Hématologie et d'Oncologie, Hôpital CHRU de Hautepierre, Strasbourg
  - Service Hématologie, Hôpital Purpan, Toulouse
  - Service Hématologie Clinique, Hôpital Bretonneau, Tours
  - Service Hématologie - Médecine Interne, Hôpitaux de Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Appelbaum FR, Gundacker H, Head DR, Slovak ML, Willman CL, Godwin JE, Anderson JE, Petersdorf SH. Age and acute myeloid leukemia. Blood. 2006 May 1;107(9):3481-5. doi: 10.1182/blood-2005-09-3724. Epub 2006 Feb 2. PMID 16455952
- [Background] Sekeres MA, Stone R. Older adults with acute myeloid leukemia. Curr Oncol Rep. 2002 Sep;4(5):403-9. doi: 10.1007/s11912-002-0034-y. PMID 12162914
- [Background] Mayer RJ, Davis RB, Schiffer CA, Berg DT, Powell BL, Schulman P, Omura GA, Moore JO, McIntyre OR, Frei E 3rd. Intensive postremission chemotherapy in adults with acute myeloid leukemia. Cancer and Leukemia Group B. N Engl J Med. 1994 Oct 6;331(14):896-903. doi: 10.1056/NEJM199410063311402. PMID 8078551
- [Background] Stone RM, Berg DT, George SL, Dodge RK, Paciucci PA, Schulman P, Lee EJ, Moore JO, Powell BL, Schiffer CA. Granulocyte-macrophage colony-stimulating factor after initial chemotherapy for elderly patients with primary acute myelogenous leukemia. Cancer and Leukemia Group B. N Engl J Med. 1995 Jun 22;332(25):1671-7. doi: 10.1056/NEJM199506223322503. PMID 7760868
- [Background] Witz F, Sadoun A, Perrin MC, Berthou C, Briere J, Cahn JY, Lioure B, Witz B, Francois S, Desablens B, Pignon B, Le Prise PY, Audhuy B, Caillot D, Casassus P, Delain M, Christian B, Tellier Z, Polin V, Hurteloup P, Harousseau JL. A placebo-controlled study of recombinant human granulocyte-macrophage colony-stimulating factor administered during and after induction treatment for de novo acute myelogenous leukemia in elderly patients. Groupe Ouest Est Leucemies Aigues Myeloblastiques (GOELAM). Blood. 1998 Apr 15;91(8):2722-30. PMID 9531581
- [Background] Pigneux A, Perreau V, Jourdan E, Vey N, Dastugue N, Huguet F, Sotto JJ, Salmi LR, Ifrah N, Reiffers J. Adding lomustine to idarubicin and cytarabine for induction chemotherapy in older patients with acute myeloid leukemia: the BGMT 95 trial results. Haematologica. 2007 Oct;92(10):1327-34. doi: 10.3324/haematol.11068. PMID 18024370
- [Background] Takagi K. [Neurophysiological and clinical aspects of autonomic centers: introduction]. Nihon Seirigaku Zasshi. 1972 May;34(5):257-61. No abstract available. Japanese. PMID 4673036
- [Background] Gardin C, Turlure P, Fagot T, Thomas X, Terre C, Contentin N, Raffoux E, de Botton S, Pautas C, Reman O, Bourhis JH, Fenaux P, Castaigne S, Michallet M, Preudhomme C, de Revel T, Bordessoule D, Dombret H. Postremission treatment of elderly patients with acute myeloid leukemia in first complete remission after intensive induction chemotherapy: results of the multicenter randomized Acute Leukemia French Association (ALFA) 9803 trial. Blood. 2007 Jun 15;109(12):5129-35. doi: 10.1182/blood-2007-02-069666. Epub 2007 Mar 6. PMID 17341661
- [Background] Hegenbart U, Niederwieser D, Sandmaier BM, Maris MB, Shizuru JA, Greinix H, Cordonnier C, Rio B, Gratwohl A, Lange T, Al-Ali H, Storer B, Maloney D, McSweeney P, Chauncey T, Agura E, Bruno B, Maziarz RT, Petersen F, Storb R. Treatment for acute myelogenous leukemia by low-dose, total-body, irradiation-based conditioning and hematopoietic cell transplantation from related and unrelated donors. J Clin Oncol. 2006 Jan 20;24(3):444-53. doi: 10.1200/JCO.2005.03.1765. Epub 2005 Dec 12. PMID 16344316
- [Derived] Largeaud L, Cornillet-Lefebvre P, Hamel JF, Dumas PY, Prade N, Dufrechou S, Plenecassagnes J, Luquet I, Blanchet O, Banos A, Bene MC, Bernard M, Bertoli S, Bonmati C, Fornecker LM, Guieze R, Haddaoui L, Hunault M, Ianotto JC, Jourdan E, Ojeda M, Peterlin P, Vey N, Zerazhi H, Yosr H, Mineur A, Cahn JY, Ifrah N, Recher C, Pigneux A, Delabesse E; French Innovative Leukemia Organization (FILO). Lomustine is beneficial to older AML with ELN2017 adverse risk profile and intermediate karyotype: a FILO study. Leukemia. 2021 May;35(5):1291-1300. doi: 10.1038/s41375-020-01031-1. Epub 2020 Sep 18. PMID 32943750